CLINICAL TRIAL: NCT02859051
Title: Efficacy of a Preparation Intervention for the Management of Children's Pain and Fear During Induction: Help From a Robot Named MEDi
Brief Title: MEDi Robot for Pain Management at Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Principal Investigator, Tanya Beran, Professor, University of Calgary
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REB16-0148
Record Dates: First submitted 2016-07-28; First posted 2016-08-08 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Cognitive Therapy
Keywords: Cognitive Behavioral Support provided by Robot

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): No intervention
- robot (Experimental): Humanoid robot interacts with child, teaching breathing and coping strategies.
  Interventions: Device: Humanoid Robot MEDi

INTERVENTIONS:
Device: Humanoid Robot MEDi — Humanoid robot programmed with cognitive-behavioral interventions such as role modeling, teaching coping strategies, positive reinforcement, parent encouragement
  Arms: robot

SUMMARY:
The purpose of this study is to determine if a preparation teaching intervention before IV insertion, taught by MEDi to children and their parents, will lead to lower levels of expected and experienced pain and fear and less distressing pain memories, as compared to children who receive standard care. In addition, it will be examined whether this preparation intervention will lead to greater parental self-efficacy, less anxiety, and less distressing pain memories as compared to controls.

DETAILED DESCRIPTION:
The primary aim is to determine the impact of using a humanoid robot in comparison to standard care. This proposal describes the first study in the world to test such novel technology for preparation teaching intervention before IV insertion. This work builds on previous research conducted by the research team and represents a logical next step for this collaborative group. This project team includes established and emerging leaders in pain management research. This will ensure successful implementation and completion of the project. These methods of teaching preparation have the potential for widespread application to other medical procedures and clinical settings (eg. oncology dentistry) and lead to improved health outcomes for children by easing their suffering and improving the quality of their healthcare encounters.

1.2 Research Questions

Research Question 1.) Does preparation administered by a humanoid robot (MEDi) reduce expectancies and experience of pain and fear of IV insertion in children?

Hypothesis 1.) Children who receive preparation by MEDi will report expecting and experiencing lower levels of fear and pain at IV insertion as compared to youth receiving standard care.

Research Question 2.) Does preparation administered by MEDi lead to higher self-efficacy and lower anxiety in parents of children undergoing IV insertion?

Hypothesis 2.) Parents of children who receive preparation by MEDi will report higher levels of self-efficacy and lower anxiety at their children's IV insertion as compared to youth receiving standard care.

Research Question 3.) Do children who receive preparation administered by MEDi and their parents have more accurate and positively estimated memories of pain and fear as compared to youth receiving standard care and their parents?

Hypothesis 3.) Children who receive preparation administered by MEDi and their parents will report more accurate and positively estimated memories of pain and fear as compared to youth receiving standard care and their parents.

Research Question 4.) Do children who receive preparation administered by MEDi prior to IV insertion and their parents expect to experience less pain, fear, anxiety, and higher self-efficacy in pain coping at future needle procedures as compared to youth receiving standard care and their parents?

Hypothesis 4.) Children who receive preparation administered by MEDi prior to IV insertion and their parents will report expecting to experience lower pain, fear, and anxiety and higher self-efficacy in pain coping at future needle procedures as compared to youth receiving standard care and their parents.

2.1 Study Design & Setting

This study is a single-centre prospective randomized, controlled, two-armed trial: (1) humanoid robot, MEDi, provides preparation for intravenous placement; and (2) standard care. Patients will be recruited from day surgery at the Alberta Children's Hospital Calgary, AB. This study will follow the high methodological standards for reporting RCTs according to the Consolidated Standards of Reporting Trials guidelines - extension for nonpharmacological treatments and this trial will be registered with clinicaltrials.gov.

2.2. Study Population

Legal guardians and/or patients with the ability to understand the study will be asked to provide written informed consent prior to participation. Day surgery patients, between the ages of 4-12 years old who are presenting for general surgery under general anesthesia, and in the American Society of Anesthesiologists class 1 or 2, will be included.

ELIGIBILITY:
Inclusion Criteria:

* presenting for general surgery under general anesthesia, and in the American Society of Anesthesiologists class 1 or 2

Exclusion Criteria:

* patient presenting for day surgery
* patient requires an intravenous placed in day surgery unit
* patient cognitively unable to self-report pain
* patient with a hearing or visual impairment or developmental disability that precludes self-reporting ability
* family or child that is unable to communicate in English
* previous allergic reaction to propofol or lidocaine

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 137 (Estimated)
Dates: Start 2016-07-08 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

PRIMARY OUTCOMES:
child's pain | at moment of child's IV start
  Faces Pain Scale-Revised (FPS-R) (Hicks, 2001)

SECONDARY OUTCOMES:
child's fear | at the moment of OR entry
  Children's Fear Scale (McMurtry, Noel, Chambers, & McGrath, 2011)
parent self-efficacy | 30 mins to 3 hours before induction
  use 0-10 numerical rating scales to report the degree to which they feel self-efficacy in their ability to help their child manage their pain and fear
parent anxiety | 30 mins to 3 hours before induction
  Parents will be asked to report on their own level of anxiety during the needle procedure using a 0-10 NRS ranging from 0 ('not at all nervous or anxious') to 10 ('most nervous or anxious').
children's memory | 2 weeks after child's induction
  , parents and children will be asked to provide their free recall of each of those periods using open-ended prompts
parents' memory | 2 weeks after child's induction
  , parents and children will be asked to provide their free recall of each of those periods using open-ended prompts

CONTACTS AND LOCATIONS:
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No